CLINICAL TRIAL: NCT04121598
Title: Project TEACH: Investigation of Momentary, Prospective Associations Between Working Memory and Eating Behavior in Children
Brief Title: Project TEACH: The Eating, Affect, and Cognitive Health Study
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: The Miriam Hospital (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Andrea Goldschmidt, Associate Professor, University of Pittsburgh
Other Study IDs: STUDY21070036; R03DK117198 (NIH)
Record Dates: First submitted 2019-10-03; First posted 2019-10-10 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Pediatric Obesity; Binge Eating
Keywords: Working Memory; Executive Functioning; Loss of Control Eating
MeSH Terms: conditions — Pediatric Obesity; Bulimia | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal Weight Control: Adolescents with a BMI percentile under 85%.
  Interventions: Other: Observational
- Overweight/Obese Control: Adolescents with a BMI percentile at 85% or higher.
  Interventions: Other: Observational
- Overweight/Obese Experimental: Adolescents with a BMI percentile at 85% or higher, who report loss of control eating episodes.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Observational data will be obtained through self-report measures, parental report measures, cognitive assessments, and a semi-structured interview.

SUMMARY:
Specific aims are to:

1. Assess variability in performance on state-level measures of working memory (WM) delivered via Ecological Momentary Assessment (EMA). The investigators expect WM performance to vary over the course of a day across participants, and to be poorer and more variable among youth with overweight/obesity and loss of control (LOC) eating relative to overweight/obese and non-overweight controls.
2. Investigate the relationship between state WM and eating behavior. The investigators expect that poorer momentary WM will predict an increased likelihood of LOC eating as assessed via EMA, and greater energy intake and poorer dietary quality as assessed via dietary recall, across participants. The investigators expect these effects to be strongest among youth with concomitant overweight/obesity and LOC eating.

DETAILED DESCRIPTION:
Pediatric overweight and obesity continue to represent major threats to public health. One cause is loss of control (LOC) eating, which involves a sense that one cannot control what or how much one is eating, affects up to 30% of youth with overweight/obesity, and may undermine weight control attempts via increased psychiatric distress, including onset of full-syndrome eating disorders. One methodology to explore factors underlying LOC eating is ecological momentary assessment (EMA), which enable examination of "in the moment" processes related to eating behavior. A neurocognitive factor implicated in LOC eating is executive functioning (EF; i.e., the ability to adaptively engage in ongoing, goal-oriented behavior). It is critical to understand the role of EF in the development of LOC eating because EF informs one's ability to understand and respond to emotions, and to engage in healthy weight regulation behaviors. In particular, working memory (WM), conceptualized as the ability to retain goal-relevant information when faced with distracting or irrelevant information, may impact regulation of eating behavior including vulnerability to LOC eating. Although WM is typically conceptualized as a trait-level factor, it is known to vary at the state-level as well, which may increase susceptibility for engaging in goal-incompatible behaviors. The proposed study uses EMA to characterize state-level WM and eating behavior in youth with overweight/obesity and LOC eating to understand how WM variations between- and within-subjects influence acute maladaptive eating. Participants will be 50 children, ages 10-17, 20 of whom are overweight/obese and report LOC eating (i.e., at least 3 objectively or subjectively large LOC episodes in the past 3 months), 20 of whom who will serve as overweight/obese controls with no LOC eating, and 10 of whom are normal-weight controls with no LOC eating.

ELIGIBILITY:
Inclusion Criteria:

* Are between the ages of 10 and 17

Exclusion Criteria:

* Are currently taking any medications known to affect weight or appetite
* Report current or past medical or psychiatric conditions known to significantly affect eating or weight (e.g., diabetes, bulimia nervosa), with the exception of binge eating disorder
* Have an Intelligence Quotient (IQ) in the borderline range or lower, or any condition affecting executive functioning (e.g., recent concussion, history of traumatic brain injury);
* Are unable to read or comprehend study materials
* Are receiving concurrent treatment for overweight/obesity

Ages: 10 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: Participants will be 50 children, ages 10-17, 20 of whom are overweight/obese and report LOC eating (i.e., at least 3 objectively or subjectively large LOC episodes in the past 3 months), 20 of whom who will serve as overweight/obese controls with no LOC eating, and 10 of whom are normal-weight controls with no LOC eating.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
BMI (Body Mass Index) | Visit 1 (pre-EMA)
  BMI will be assessed using height and weight (cm/g)
Eating Behavior | Visit 1 (pre-EMA)
  Eating behavior will be assessed using the Eating Disorder Examination (EDE), a semi-structured interview. Global scores are calculated, with higher scores indicating higher disordered eating symptomology.
Eating Behavior | Across 2-week EMA period
  Eating behavior will be assessed through Nutritional Data System for Research (NDSR) software, which calculates daily macro-nutrient numbers based on self-report food recalls.
Working Memory | Visit 1 (pre-EMA)
  Working memory will be assessed using 3 NIH Toolbox measures: the list sort task, the Flanker task, and the dimensional card task.
Working Memory | Across 2-week EMA period
  Working memory will be assessed using a number changing task created for the purpose of this study. Sum correct responses will be scored with higher scores indicating a higher number of correct responses.
Spatial Reasoning | Across 2-week EMA period
  Spatial reasoning will be assessed using a moving grid task created for the purpose of this study. Sum correct responses will be scored with higher scores indicating a higher number of correct responses.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea B. Goldschmidt, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- Weight Control & Diabetes Research Center, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-07-10): https://cdn.clinicaltrials.gov/large-docs/98/NCT04121598/ICF_000.pdf